CLINICAL TRIAL: NCT05207176
Title: An Open-label, Single-center, Parallel, Single and Multiple Oral Dose Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of DWP16001 in Healthy Koreans, Caucasians, and Hispanics
Brief Title: Study to Evaluate the Safety and PK Properties of DWP16001 in Healthy Subjects With Various Ethnicities
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWP16001107
Record Dates: First submitted 2022-01-12; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2021-11

CONDITIONS: Healthy
MeSH Terms: interventions — Enavogliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DWP16001 (Experimental): Total number of subjects: 24 (8 Korean, 8 Caucasian, and 8 Hispanic)
  Interventions: Drug: DWP16001

INTERVENTIONS:
Drug: DWP16001 — Subjects should fast except for drinking water after 10 p.m. in order to maintain a fasting state for at least 10 hours before administration. On dosing days (5d to 10d), except for 1d and 11d, breakfast can be consumed from about 1 hour after administration of the clinical trial drug. Subjects should swallow the investigational drug whole with 150 mL of water, and should not chew the drug before swallowing. Subjects should fast for 4 hours after dosing, and can drink water freely from 2 hours after dosing.

SUMMARY:
An open label, single center, parallel, single and multiple oral dose study to evaluate the pharmacokinetics, pharmacodynamics, safety and tolerability of DWP16001 in healthy Koreans, Caucasians, and Hispanics

DETAILED DESCRIPTION:
This study is conducted with single center, parallel design, single and repeated administration and repeated administration.

1. Screening (28d~ 2d) For volunteers, screening tests such as questionnaire, physical examination and clinical examination are conducted within 4 weeks (-28d~-2d) from the date of administration of the clinical investigational drug (1d), and subjects judged to be suitable for this clinical trial are selected.
2. Dosing and Pharmacokinetics/Pharmacodynamic Evaluators (1d to 12d) The subjects who are judged to be suitable for this clinical trial are admitted to the clinical trial center of Seoul National University Hospital in the afternoon of 1 day (-1d) before administration. In order to maintain an empty stomach for at least 10 hours before administration of clinical trial drugs, fast except for drinking water after 10 p.m.
3. PSV (17d ~ 21d) The post-study visit is conducted on 17d to 21d, about one week after the last dosing date.

ELIGIBILITY:
Inclusion Criteria:

1. A healthy adult between 19 and 50 years of age at the time of screening 2. Koreans, Caucasian, and Hispanics are classified according to the following criteria.

1. Korean: A Korean ethnic group born in Korea or outside Korea who has lived abroad for 10 years and has Korean parents and grandparents.
2. Caucasian: Born in Europe, living abroad in Europe for 10 years, Europeans with European parents and grandparents
3. Hispanic: Subjects of Latin American races with parents and grandparents who are Latin American, having nationalities from Mexico, Puerto Rico, Cuba, Latin America, or other Spanish cultures.

3. At the time of screening test, if the weight is more than 50.0 kg or less than 90.0 kg, the body mass index (BMI) is 18.0 kg/m^2 or more 30.0 kg/m^2 or less (*body mass index, kg /m^2) = weight (kg) / [height (m)] 2) 4. In the case of female volunteers, factors such as not necessarily pregnant or lactating or surgical infertility (both difficulty tube closure, hysterectomy, both difficulty tube resection, both ovarian resection, etc.) 5. A person who has heard sufficient explanation of this clinical trial and fully understood it, voluntarily decided to participate, and agreed in writing to comply with precautions.

Exclusion Criteria:

1. Clinically significant hepatometer (severe liver disorder, etc.), kidney (severe renal disorder, etc.), nervous system, immune system, respiratory system, digestive system, endocrine system, blood • tumor, cardiovascular system (heart failure, Torsades de points, etc.), urinary system, mental system, etc.
2. A person who has a history of hypersensitivity or clinically significant hypersensitivity to DWP16001 and other drugs (aspirin, antibiotics, etc.), including homogeneous drugs.
3. Those with a history of gastrointestinal diseases (gastrointestinal ulcers, gastritis, stomach cramps, gastroesophageal reflux disease, Crohn's disease, etc.) or surgery that may affect the safety and pharmacokinetic/pharmacodynamic evaluation of DWP16001 (however, simple appendicectomy, excluding hernia surgery)
4. The person who showed the following results in the screening test. 1) Blood AST (SGOT), ALT (SGPT):> Upper limit of normal range × 1.5 2) Creatine cleaning rate calculated through MDRD equation: <90 mL/min 3) Serum glucose on an empty stomach: >110 mg/dL or <70 mg/dL 4) Serum test (syphilis test, hepatitis B test, hepatitis C test, human immunodeficiency virus (HIV) test) results are positive factors.
5. Those with a systolic blood pressure <90 mmHg or >150 mmHg or diastolic blood pressure <60 mmHg or >100 mmHg in vital signs measured in the sitting position after resting for more than 3 minutes
6. Those who have a history of drug abuse or who have tested positive for drugs of abuse in urine screening tests
7. Those who have taken any prescription drugs or herbal medicines within 2 weeks before the expected first dose, or have taken any over-the-counter (OTC) drugs, health functional foods, or vitamins within 1 week (however, different conditions according to the judgment of the researcher) In this reasonable case, you can participate in the clinical trial) or those who are expected to take it
8. Those who have taken drugs that induce or inhibit drug metabolizing enzymes, such as barbiturates, within 1 month before the expected first administration date
9. A person who participated in other clinical trials (including biological equivalence tests) and administered drugs for clinical trials within 6 months of the expected first dose date.
10. A person who donated whole blood within 2 months prior to the expected first dose or donated ingredients within 1 month prior to the expected first dose date, or received a blood transfusion within 1 month prior to the expected first dose date.
11. A person who is unable to drink continuously (exceeds 21 units/week, 1 unit = 10 g of pure alcohol) or to abstain from drinking during the period from 3 days before the expected first administration date to the last discharge.
12. A current smoker (however, if he/she quit smoking three months before the expected first dose date, he/she can be selected as a test subject) or a person who cannot stop smoking during the period from the time of discharge.
13. Those who cannot refrain from eating grapefruit (grapefruit)-containing food during the period from 3 days before the expected first administration date to the last discharge
14. A person who continuously consumed excessive caffeine (> 5 units/day) or who cannot prohibit the intake of caffeine/caffeine-containing foods (coffee, tea (black tea, green tea, etc.), soda, coffee milk, nutritional tonic drinks, etc.) during the expected first 3 days to the last discharge.
15. Those who cannot use an appropriate double contraceptive method or medically acceptable method of contraception for themselves, their spouse, or their partner during the entire clinical trial period, and those who do not agree not to donate sperm or eggs until the relevant period

    * Medically acceptable contraceptive method

      1. The use of intrauterine devices with proven pregnancy failure rates in oneself or spouse (or partner)
      2. Use of both blocking contraception method (for men or women) and skin killer at the same time.
      3. Surgery of the person or partner (vascularization, arthroplasty/ligation, hysterectomy
16. Those who do not meet the above selection criteria or who are judged by the researcher as unsuitable to participate in the clinical trial due to reasons other than those that fall under the exclusion criteria

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-02-14 (Estimated); Primary Completion 2022-04-08 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Cmax | Single dose: 0 (pre-dose), 0.25 to 96 hours post dose on Day 1, Multi-dose: 0 (pre-dose), 0.25 to 24 hours post dose on Day 11
  Cmax of plasma DWP16001
AUClast | Single dose: 0 (pre-dose), 0.25 to 96 hours post dose on Day 1, Multi-dose: 0 (pre-dose), 0.25 to 24 hours post dose on Day 11
  AUClast of plasma DWP16001